CLINICAL TRIAL: NCT03028259
Title: Does Plasma Glucose Variability in Obese Diabetic Pregnancies Influence Maternal or Neonatal Outcomes?
Brief Title: Glucose Variability
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Laura Vricella, MD, PI, St. Louis University
Other Study IDs: 24669
Record Dates: First submitted 2017-01-10; First posted 2017-01-23 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Glucose Variability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lab results: monitoring of
  Interventions: Other: lab results

INTERVENTIONS:
Other: lab results — Comparison of lab results

SUMMARY:
A retrospective data review of 243 pregnant women (≤32 wks gestational age), dtat collected prior to 5/18/2014, with GDM, or T2DM, and their infants (until discharge from the hospital, typically up to 1 week after deliver) will be conducted. These women are of any age and all ethnic backgrounds delivering at St. Mary's Health Center.

DETAILED DESCRIPTION:
Maternal glucose control is considered to be a major determinant of neonatal outcome in pregnancies complicated by diabetes. Studies have examined the link between neonatal mortality and morbidity using specific mean preprandial or postprandial plasma glucose levels, however, have not taken into account the daily wide excursions that occur in maternal glucose levels. Limited data are available on glucose variability (GV) in pregnancy and affect on maternal or neonatal outcomes. A recent study amongst diabetics showed that glucose variability between two data points, a morning fasting blood glucose and an afternoon blood glucose, increased the rate of adverse neonatal outcomes1. Glycosylated hemoglobin (A1c), which has been considered the "gold standard" for diabetes control since the Diabetes Control and Complication Trial (DCCT)2, lacks the specificity to predict pregnancy outcomes. Through review of data, we propose to examine other methods of evaluating daily maternal glucose variations to determine the correlation to maternal and neonatal outcomes.

The objective of this study is to determine the effect of glucose variability and/ or other elements on maternal and neonatal outcomes in the obese diabetic patient. We hypothesize that glucose variability will be a stronger indicator of neonatal outcome than A1c or any single given blood glucose value. Glucose variability, including the magnitude of hyperglycemia or the incidence of acute maternal hypo- or hyperglycemic events, will be explored. We hypothesise that obese pregnant women with higher magnitude of glucose fluctuations have more maternal and fetal co morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Women with diabetes in pregnancy of any age, any ethnic background who deliver at St. Mary's Health Center, 1/1/2000 to 5/18/2014.

Exclusion Criteria:

* Data collected ager 5/18/2014

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women with diabetes in pregnancy of any age, any ethnic background
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2014-06-24 (Actual)

PRIMARY OUTCOMES:
glucose levels | 1 year
  the effect of glucose variability on maternal and neonatal outcomes in the obese diabetic patient.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vricella, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No